CLINICAL TRIAL: NCT02898688
Title: A Comprehensive Pre-Natal Intervention to Increase Vaccine Coverage (P3+): Practice, Provider, Patient Level Interventions
Brief Title: P3+ Intervention Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Robert Bednarczyk, Assistant Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00090267; 5R01AI110482-02 (NIH)
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Vaccination
Keywords: Influenza vaccine; Pertussis vaccine; Perinatal vaccination; Infant vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Site + Control Patient (Other): The obstetric practice site is randomized to be a control site and the patient is randomized to the control group.
  Interventions: Behavioral: Control Site; Behavioral: Patient-level Control Group
- Control Site + Intervention Patient (Experimental): The obstetric practice site is randomized to be a control site and the patient is randomized to receive the intervention.
  Interventions: Behavioral: Control Site; Behavioral: Patient-level Intervention Group
- Intervention Site + Control Patient (Experimental): The obstetric practice site is randomized to be an intervention site and the patient is randomized to the control group.
  Interventions: Behavioral: Intervention Site; Behavioral: Patient-level Control Group
- Intervention Site + Intervention Patient (Experimental): The obstetric practice site is randomized to be an intervention site and the patient is randomized to receive the intervention.
  Interventions: Behavioral: Intervention Site; Behavioral: Patient-level Intervention Group

INTERVENTIONS:
Behavioral: Control Site — Control sites will continue with their standard practice regarding discussing vaccines with their patients.
  Other Names: Practice/provider-Level Control
  Arms: Control Site + Control Patient; Control Site + Intervention Patient
Behavioral: Intervention Site — Intervention Sites will each assign a Vaccine Champion and will have Assessment, Feedback, Incentives, and eXchange (AFIX) visits. AFIX is a quality improvement program to raise immunization coverage levels, reduce missed opportunities to vaccinate, and improve standards of practices at the provider level. A Continuing Medical Education (CME) module will be given to all providers, covering the recommended maternal vaccinations and how to talk to patients about vaccines. Intervention sites will have access to written materials covering all recommended maternal and infant vaccinations, the diseases they prevent, potential adverse reactions and common patient questions with talking points and references for each topic.
  Other Names: Practice/provider-Level Intervention
  Arms: Intervention Site + Control Patient; Intervention Site + Intervention Patient
Behavioral: Patient-level Control Group — Participants randomized the control arm will complete a computer-based questionnaire, on an iPad with a preloaded app. The questionnaire asks about vaccine knowledge, attitudes, and beliefs and the participant's intent to receive vaccinations during pregnancy and to vaccinate their baby. The questionnaire includes questions requiring a "yes" or "no" response, degree of agreement with vaccine-related statements (ranging from strongly agree to strongly disagree), questions to capture the vaccines participants plan to get for themselves and their children, and open-ended questions.
  Arms: Control Site + Control Patient; Intervention Site + Control Patient
Behavioral: Patient-level Intervention Group — Participants randomized to the intervention arm will complete a computer-based questionnaire on an iPad with a preloaded app, prior to watching informational videos covering topics on maternal and childhood vaccines. The questionnaire asks about vaccine knowledge, attitudes, beliefs, and the participant's intent to receive vaccinations during pregnancy and to vaccinate their baby. The questions require "yes" or "no" responses, degree of agreement with vaccine-related statements (ranging from strongly agree to strongly disagree), and open-ended responses. After watching at least one informational video, the participant completes a questionnaire asking about the perceived usefulness of the app, degree of agreement with the vaccine information presented in the video, and ways to make the app more useful to participants.
  Arms: Control Site + Intervention Patient; Intervention Site + Intervention Patient

SUMMARY:
This study will address vaccine uptake both for pregnant women and for their children, through 20 months of age, to test the hypothesis that exposure to the P3+ intervention package will increase the likelihood a pregnant woman gets herself vaccinated against influenza and pertussis before delivery and get her child vaccinated on time. This study builds off of a prior intervention, developed by Emory, at the practice, provider, and patient levels (P3) to develop, implement and evaluate an enhanced intervention (P3+) to improve vaccination uptake among pregnant women, and later, their children.

DETAILED DESCRIPTION:
This study will address vaccine uptake both for pregnant women and for their children, through 20 months of age, to test the hypothesis that exposure to the P3+ intervention package will increase the likelihood a pregnant woman gets herself vaccinated against influenza and pertussis before delivery and get her child vaccinated on time.

This study uses a multi-level factorial design which randomizes at both the practice and the patient level. Obstetric practices in Georgia and Colorado will be randomized to be either an intervention practice or a control practice. The women recruited in the practices and enrolled in the study will be randomly assigned to the intervention arm or the control arm.

Women randomized to the intervention arm will complete a computer-based questionnaire (administered via iPad with a preloaded study app) which asks for their basic demographic and contact information and asks questions about their vaccine knowledge, attitudes, and beliefs. Immediately following the questionnaire, participants will receive the individual level intervention (videos providing information on vaccines) on the same iPad. In order to best answer their questions and not provide information beyond the scope of what the study participants need or want, the videos provided to each participant will be selected based on responses to the survey questions. There are 6 videos: one discusses the dangers of the diseases prevented by vaccines, and the others address specific vaccine concerns (concerns include vaccine ingredients, children receiving simultaneous vaccines (multiple vaccines at one time), and the safety of receiving the tdap or flu vaccine during pregnancy). If the participant does not have any concerns, they will only see the video about dangers of vaccine preventable diseases. Participants expressing concerns in the survey will receive up to two videos addressing those concerns, based on an order of priority determined by the study researchers.

Women randomized to the control arm will also complete a computer-based questionnaire which includes their personal information and vaccine knowledge, attitudes, and beliefs questions but will then continue to receive usual prenatal care rather than view informational videos.

All enrolled women complete two follow-up surveys when their children are 30 days and 18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Have not previously participated in this study
* Currently pregnant
* Up to 26 weeks gestational age
* Able to understand and communicate in English

Exclusion Criteria:

* Have received pertussis vaccine during the current pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2200 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Number of women receiving influenza vaccination | Up to 34 weeks
  Whether or not the participant chose to receive the flu vaccine during pregnancy (between the baseline visit and birth of infant) will be compared between study arms
Number of women receiving pertussis vaccination | Up to 34 weeks
  Whether or not the participant chose to receive the pertussis vaccine during pregnancy (between the baseline visit and birth of infant) will be compared between study arms
Timely childhood vaccinations | 20 months
  Childhood vaccination will be assessed as timely uptake of childhood vaccines by calculating average days under-vaccinated. The total number of days under-vaccinated will be divided by the number of vaccines a child should have received, according to the Advisory Committee on Immunization Practices (ACIP) schedule, to give the average number of days under-vaccinated across all recommended vaccines. This can range from 0 to 415 days in the first 20 months of life. The average number of days under-vaccinated will be modeled as a continuous variable, and the distribution of days under-vaccinated will be evaluated, in total and by vaccine where possible, to identify specific patterns of interest for follow-up.

SECONDARY OUTCOMES:
Changes in maternal vaccine knowledge | Up to 106 weeks (baseline visit until 18 months post delivery)
  Maternal vaccine knowledge will be collected by the app surveys at different time periods, including before receiving the patient-level intervention, immediately after receiving the intervention, and 30 days and 18 months after the birth of the child. The survey questions assessing these outcomes will most often be measured on a Likert scale. Changes in these outcomes over time will be compared between mothers in the different study arms.
Changes in maternal vaccine attitudes | Up to 106 weeks (baseline visit until 18 months post delivery)
  Maternal vaccine attitudes will be collected by the app surveys at different time periods, including before receiving the patient-level intervention, immediately after receiving the intervention, and 30 days and 18 months after the birth of the child. The survey questions assessing these outcomes will most often be measured on a Likert scale. Changes in these outcomes over time will be compared between mothers in the different study arms.
Changes in maternal vaccine beliefs | Up to 106 weeks (baseline visit until 18 months post delivery)
  Maternal vaccine beliefs will be collected by the app surveys at different time periods, including before receiving the patient-level intervention, immediately after receiving the intervention, and 30 days and 18 months after the birth of the child. The survey questions assessing these outcomes will most often be measured on a Likert scale. Changes in these outcomes over time will be compared between mothers in the different study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bednarczyk, PhD, Principal Investigator — Emory University; Daniel Salmon, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (23):
- United States (23):
  - CU Center for Midwifery, Aurora, Colorado
  - CU Maternal and Fetal Medicine Clinic, Aurora, Colorado
  - University Nurse Midwives, Aurora, Colorado
  - Boulder Women's Care, Boulder, Colorado
  - St. Joe's Midwives, Denver, Colorado
  - Partners in Women's Health at Rose, Denver, Colorado
  - Rocky Mountain OBGYN, Denver, Colorado
  - Colorado Mountain Medical, Edwards, Colorado
  - Bella Natural Women's Care, Englewood, Colorado
  - Associates in Women's Health, Golden, Colorado
  - Women's Health Group Thornton, Thornton, Colorado
  - Atlanta Women's Specialists, Alpharetta, Georgia
  - Roswell Ob/Gyn, Alpharetta, Georgia
  - Athens Midwifery, Athens, Georgia
  - Athens Ob-Gyn, Athens, Georgia
  - Women's Healthcare Associates of Athens, Athens, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Riverbend OB/GYN and Counseling, Atlanta, Georgia
  - Peachtree Women's Clinic, Cumming, Georgia
  - Comprehensive Women's OB/GYN, Duluth, Georgia
  - Dunwoody Ob-Gyn, Dunwoody, Georgia
  - Atlanta Gynecology & Obstetrics, Lilburn, Georgia
  - Women's Medical Center, Tyrone, Georgia

REFERENCES:
- [Derived] Dudley MZ, Omer SB, O'Leary ST, Limaye RJ, Ellingson MK, Spina CI, Brewer SE, Bednarczyk RA, Chamberlain AT, Malik F, Frew PM, Church-Balin C, Riley LE, Ault KA, Orenstein WA, Halsey NA, Salmon DA. MomsTalkShots, tailored educational app, improves vaccine attitudes: a randomized controlled trial. BMC Public Health. 2022 Nov 21;22(1):2134. doi: 10.1186/s12889-022-14498-7. PMID 36411403
- [Derived] Dudley MZ, Limaye RJ, Omer SB, O'Leary ST, Ellingson MK, Spina CI, Brewer SE, Chamberlain AT, Bednarczyk RA, Malik F, Frew PM, Salmon DA. Factors associated with referring close contacts to an app with individually-tailored vaccine information. Vaccine. 2020 Mar 17;38(13):2827-2832. doi: 10.1016/j.vaccine.2020.02.019. Epub 2020 Feb 22. PMID 32098739

DOCUMENTS (1):
  • Informed Consent Form (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT02898688/ICF_000.pdf